CLINICAL TRIAL: NCT06810193
Title: Monitoring & Mitigation of Neurologic Injuries to Optimize Resilience After Repetitive Head Impacts
Acronym: MONITOR-RHI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jeffrey Bazarian, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00010101; US Department of Defense (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2025-01-25; First posted 2025-02-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Head Injuries
Keywords: Repetitive Head Impacts
MeSH Terms: conditions — Craniocerebral Trauma | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational (Ad-Lib Exercise) Arm (No Intervention): All participants will undergo neurologic outcome testing with optical coherence tomography/angiography (OCT/A) at pre- and post-season and 2 weeks after the end of the season. For two weeks at the end of the sport season, participants will be instructed to refrain from sports involving head contact but to otherwise exercise ad-lib.
- Intervention (Exercise or Stretching) Arm (Experimental): Athletes and athlete cadets will be administered OCT/A and a novel neurologic test battery at pre- and post-season, and 2 weeks after the end of the season. After the end-of-season assessments, participants will be randomized to 2 weeks of either 30 minutes of daily aerobic exercise or to 30-minutes of prescribed stretching.
  Interventions: Other: Aerobic exercise

INTERVENTIONS:
Other: Aerobic exercise — After the end-of-season assessments, participants in the Intervention (Exercise or Stretching) arm will be randomized to 2 weeks of daily aerobic exercise for 30 minutes or to 30-minutes of prescribed stretching.
  Arms: Intervention (Exercise or Stretching) Arm

SUMMARY:
The purpose of this Phase 2, double-arm study is to identify repetitive, non-concussive head impacts that impair neurologic functioning, and to test treatments that can mitigate these effects and return functioning to normal as quickly as possible.

DETAILED DESCRIPTION:
Up to 350 total collegiate athletes and athlete-cadets will be enrolled. Approximately 290 participants participating in varsity contact sports (e.g. soccer, football, etc.) at colleges/universities or military colleges, and up to 60 non-contact athletes/cadets participating in non-contact varsity sports (e.g. swimming, tennis, etc.) will be recruited as controls for the Observational arm; approximately half the participants will be female.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Collegiate athlete or athlete-cadet anticipated to be an active member of a varsity sport team.

Exclusion Criteria:

* Any head, neck, or face injury in the 3 months prior to enrollment that precludes participation in contact sports or wearing a mouth guard sensor
* History of neurological or psychiatric disorders or neurological disorders that impact electrical activity in the brain (such as seizure disorders), or diagnosed learning disability, that in the opinion of the investigator, would interfere with participation in the study.
* Participants currently undergoing active treatment for migraine, depression and/or anxiety or ADHD will not be excluded as these are high prevalence conditions in the adolescent and collegiate population (8-30%). However, exploratory stratified analyses will be conducted where possible.
* Participants with eye conditions or diseases that could impact the blood vessels in the eye.
* Determination that the participant is unsuitable for study entry or potentially unable to complete all aspects of the study based on the judgement of the Site Investigator or Study PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Optical Coherence Tomography (OCT) of Cerebrospinal Fluid Thickness in the Macula (Part of the Retina) | Pre-season and post-season, 2 weeks
  A primary OCT variables examined will be macula cerebrospinal fluid (CSF) thickness (an indicator of the gain or loss of neurons or glia in the inner nuclear, ganglion cell and nerve fiber layer).
Change in Blood Serum Concentrations of Glial Fibrillary Acidic Protein (GFAP) | Baseline 4 to 7 months
  Glial Fibrillary Acidic Protein (GFAP) concentration will determine if there is a 11.9 pg/mL or greater change in GFAP in each participant over the course of the study.
Change in Blood Serum Concentration of Neurofilament light chain (NfL) in a blood sample | Baseline 4 to 7 months
  The neurologic test battery consists of blood draws for serum brain proteins: Neurofilament light chain (NfL) concentrations will be observed for changes over the course of the study.
Change in p-231Tau serum concentration in a blood sample | Baseline 4 to 7 months
  The neurologic test battery consists of blood draws for serum brain proteins: p231Tau will be observed for changes over the course of the study.
Change in Concussion Index as measured with Quantitative Electroencephalogram (qEEG) | Baseline 4 to 7 months
  The Quantitative Electroencephalogram (qEEG) Concussion Index (CI) includes measures of power (absolute and relative), mean frequency, connectivity (asymmetry, coherence, phase lag, phase synchrony), complexity (fractal dimension and scale-free activity), and information theory (entropy), across and within frequency bands.
Change in near-point convergence (NPC) | Baseline 4 to 7 months
  Near point of convergence (NPC) is a measurement of how close an object can be brought to the eyes while the eyes are focused on it.
Change in Choice reaction time (CRT) | Baseline 4 to 7 months
  Choice reaction time (CRT) refers to the time it takes for a person to react to a stimulus by selecting a specific response from multiple options.
Change in blink reflex test | Baseline 4 to 7 months
  A blink reflex test, also known as a corneal reflex test, is a non-invasive procedure that measures the electrical activity of the facial nerves when stimulated.
Optical Coherence Tomography (OCT) to detect signs of neurodegenertaion in the Retina | Pre-season and post-season, 2 weeks
  OCT will be used to measure the cup-to-disc ratio of the optic disc, and indicator of neurodegeneration.
Optical Coherence Tomography/Angiography (OCT/A) to assess the vascular structure in the retina | Pre-season and post-season, 2 weeks
  Retinal vascular structure will be acquired using the OCT angiography (OCT/A). The primary OCT/A variable examined will be foveal avascular zone (FAZ) area reflecting the size of the central portion of the macula which contains no blood vessels, and which increases in size with loss of capillaries in the surrounding region).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University at Buffalo, Amherst, New York
  - University of Rochester, Rochester, New York
  - The Citadel, The Military College of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No